CLINICAL TRIAL: NCT01707758
Title: Detection of Cancer-Specific Active Proteases in Blood Via Fluorescence
Status: Withdrawn | Type: Observational
Why Stopped: Trial terminated - Nanoscale Company out of business
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 13421
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; nanoparticle; proteases; cell survival; tumor progression; angiogenesis; tissue remodeling/invasion
MeSH Terms: conditions — Pancreatic Neoplasms; Disease Progression

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Approximately 1 tablespoon of blood will be collected from each subject.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pancreatic cancer: This study will collect blood from 36 patients with known or suspected pancreatic cancer and from 12 healthy cancer-free subjects.

SUMMARY:
The primary objective is to develop a rapid in vitro screening assay for detection of pancreatic cancer biomarkers in blood of patients with pancreatic cancer.

DETAILED DESCRIPTION:
The goal of the project is to develop a rapid in vitro screening assay for detection of cancer biomarkers in blood. The aim is testing and optimization of nanoparticle sensors, based on cyanine dyes that are chemically linked to Fe/Fe3O4 nanoparticles via protease-selective consensus (cleavage) sequences. The focus is on the quantitative determination of active cancer-specific proteases in blood via simple fluorescence measurements. The matrix metalloproteinases, urokinase-type plasminogen activator, and cathepsins, are up-regulated in the vast majority of progressing cancers and can, therefore, serve as markers for cell survival/tumor progression, angiogenesis, and tissue remodeling/invasion

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Pancreatic Cancer Patients:

* Patients will either have a histologic diagnosis of pancreatic carcinoma or a clinical picture consistent with pancreatic cancer and will be undergoing surgery or a diagnostic procedure to confirm the diagnosis.
* Patients will have had no prior treatment or surgery

Inclusion Criteria for Healthy Subjects:

* Subjects will have no prior history of any cancer

Exclusion Criteria:

Exclusion Criteria for Pancreatic Cancer Patients

* Any prior treatment for pancreatic cancer
* Poorly controlled diabetes

Exclusion Criteria for Healthy Subjects

* Poorly controlled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the University of Kansas Cancer Center prior to any treatment for their pancreatic cancer. Final histology and staging will be recorded and correlated with protease concnentration. Healthy subjects will be recruited from the University of Kansas and Kansas State community.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Williamson, MD, Principal Investigator — University of Kansas Medical Center Cancer Center